CLINICAL TRIAL: NCT06955832
Title: Early Identification of Brain Lesions in Multiple Sclerosis With Phase Sensitive Inversion Recovery MRI: A Cross-sectional Study
Brief Title: Early Identification of Brain Lesions in Multiple Sclerosis With Phase Sensitive Inversion Recovery MRI
Status: Recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmad Elsayed, Neurology Specialist, Benha University
Other Study IDs: MD 3-5-2024
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cortical lesions; MRI; Early diagnosis; McDonald criteria
MeSH Terms: conditions — Multiple Sclerosis; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to compare the diagnostic accuracy of Phase-Sensitive Inversion Recovery (PSIR) MRI versus conventional T2-weighted (T2W) and Fluid Attenuated Inversion Recovery (FLAIR) sequences in detecting early brain lesions in patients with Multiple Sclerosis (MS). The study will include male and female participants aged 15-65 years diagnosed with MS per the 2017 McDonald criteria.

This study hypothesizes that:

* PSIR MRI will detect a significantly higher number of cortical lesions (intracortical, leukocortical, and juxtacortical) compared to conventional T2W and FLAIR sequences in MS patients (p < 0.05).
* Lesions identified exclusively by PSIR will correlate more strongly with clinical measures (EDSS disability scores and SDMT cognitive performance) than those detected by T2W/FLAIR alone, suggesting PSIR's superior sensitivity to clinically relevant pathology.

DETAILED DESCRIPTION:
Introduction Multiple sclerosis (MS) is an immune, demyelinating disease that assaults myelinated axons in the central nervous system (CNS), damaging the myelin and axon to varying degrees. Inflammation, neurodegeneration, and gliosis are hallmarks of MS. Perivascular lymphocytic infiltrate and macrophages destroy the myelin sheaths that pathologically wrap neurons.

In most cases, the condition is relapsing-remitting, with brief bouts of neurologic impairment that resolve entirely. MS pathophysiology is not fully understood but may be connected to hereditary predisposition and a putative non-genetic trigger that results in a sustaining autoimmune disease leading to recurring immunological attacks on CNS.

Several risk factors lead to MS's development, including age, sex, race, heredity, geography, and infections such as herpes simplex, chlamydia, and rabies. MS is likely the result of a complicated interplay between genetics, food, and the environment. MS is primarily caused by an autoimmune attack on the CNS due to hyper immunity. Numerous postulated pathways have been proposed, but the proposed "outside-in" mechanism involves CD4+ proinflammatory T cells.

Cortical demyelinating lesions are defined as focal lesions located entirely inside of the cortical grey matter (pure cortical lesions) or extending partially towards the underlying juxtacortical white matter (leukocortical lesions). These lesions constitute a distinctive characteristic of MS, and their presence aids in identifying patients with an isolated clinical syndrome at higher risk of developing a second clinical episode and, therefore, in predicting the risk of conversion to clinically defined MS. In addition, cortical lesions are not identified in other disease processes which may mimic MS, such as migraine.

Cortical gray matter lesions are a common ﬁnding in neuropathlogical studies of multiple sclerosis (MS), and in some studies are more extensive than lesions seen in white matter. However, conventional MRI using T2-weighted, or ﬂuid-attenuated inversion recovery (FLAIR) sequences, reveals few cortical lesions, and is considerably less sensitive to cortical than white matter lesions.

Sensitive method to detect cortical lesions in vivo might assist the diagnosis of MS and provide a new way to monitor the course of MS and its medication by treatment.

Accurate detection and classification of purely intracortical lesions in multiple sclerosis (MS) are important in understanding their role in disease progression and impact on the clinical manifestations of the disease. However, detection of these lesions with conventional MR imaging remains a challenge.

Recent studies have shown that the phase-sensitive inversion recovery (PSIR) sequence, consisting of a heavily T1-weighted sequence with higher signal-to-noise ratio, intensity and gray-white matter contrast has been shown to improve Cortical Lesion detection and inversion recovery combined with phase-sensitive reconstruction, had the highest lesion-to-brain contrast and lesion-limit definition. Therefore, this sequence seemed particularly promising for the detection of cortical lesions.

Subjects and Methods

• Study Design: This study is a cross sectional study.

• Study subjects: The study will be conducted on patients with multiple sclerosis, they will be recruited from neurology department of Banha university hospitals, El Mounira MS unit and Naser specialized hospital MS unit.

• Sample size: Sample size was calculated by Stata Corp. 2021. Stata Statistical Software: Release 17. College Station, TX: Stata Corp LLC., with respect to comparing the ability of detecting cortical lesions with phase sensitive inversion recovery and conventional recovery in MS patients.

Using t test model: difference between two independent means, expected effect size of 0.8; required sample size is 30 MS patients, using α error 5% and a power of 80%.

• Study tools:

Patients with MS will be identified according to:

* Revised McDonald criteria. The "McDonald Criteria" have been extensively assessed and used since 2001 and revised in 2005 and 2017
* Expanded Disability Status Scale (EDSS):

Expanded Disability Status Scale (EDSS) is the most commonly used scale in multiple sclerosis (MS) patients. EDSS is a very effective method of reflecting disability. The EDSS provides a total score on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability.

• Symbol Digit Modalities Test (SDMT): Is one of the most widely used rapid cognition tests for adults with MS, used to evaluate the cognitive psychometric profile captured by the SDMT to identify whether different cognitive processes independently underlie performance.

* All patients will be subjected to:

  * An informed consent will be taken from every patient to confirm approval of participation in the study.
  * Complete history taking that include:

    * Personal history.
    * Past medical and past surgical history.
    * Family history.
  * Complete physical examination including:

    * General examination:
    * Local examination of the affected system.
    * Neurologic examination
  * Investigations
* Imaging:

MRI will be performed at 1.5T using an 8-channel SENSE receive-only head coil with the same protocol for both baseline and follow-up, and patients will be repositioned according to established guidelines.

All images will be analyzed off-line and inspected for presence of major artifacts.

The PSIR images will be obtained for each patient in every session as part of routine MRI sequences, which also will include conventional T2W-TSE and FLAIR., Cortical lesion that will be identified on PSIR will be compared slice by slice with those identified on FLAIRE in order to obtain a corresponding classification.

Two independent neuroradiologists separately will assess all MR images. The number of plaques will be determined in each sequence and compared blindly among sequences.

The plaques will be defined as hyperintense in T2W and FLAIR and as hypointense in PSIR.

The number of plaques will be determined in terms of IC, leukocortical (LC), and juxtacortical (JC) regions. The IC lesions are confined to the GM, while lesions that involved both the cortex and the adjacent WM are identified as LC lesions. Finally, the JC lesions will be WM lesions involving the subcortical U-fibers.

Ethical consideration:

An informed consent will be taken from all subjects prior to the imaging. Ethical considerations according to the ethical committee of Benha University. Statistical analysis All statistical analyses will be performed using Statistical Package for the Social Sciences (SPSS, Version 20.0, Chicago, Illinois). Student t and Mann Whitney tests will be used to compare numerical data. Chi square test will be used to compare categorical data. Spearman's rank correlation coefficients will be used to determine the associations between variables. All p values will be reported as two-sided significance levels and considered statistically significant when p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15-65 years.
* Both sexes.
* Patients with MS according to McDonald Criterion

Exclusion Criteria:

* Age less than 15 years old.
* Patients with stroke or previous intracranial hemorrhage.
* Contraindications to MRI scans.
* MS mimics.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll participants from three clinical sites in Egypt:
  * Neurology Department, Banha University Hospitals (Benha, Qalyubia Governorate).
  * El Mounira MS Unit (Cairo).
  * Naser Specialized Hospital MS Unit (Cairo).
  Recruitment Setting:
  * Outpatient MS clinics at all three sites
  * Inpatient neurology services at Banha University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number and classification of cortical lesions | 18 months
  Total cortical lesion count (sum of intracortical [IC], leukocortical [LC], and juxtacortical [JC] lesions) detected by each MRI sequence (PSIR vs. T2W vs. FLAIR), assessed by two independent neuroradiologists..
  Lesion subtype distribution:
  * IC lesions (confined to gray matter).
  * LC lesions (spanning gray-white matter).
  * JC lesions (subcortical U-fiber involvement).

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Banha University Hospitals, Banhā, Qalyubia Governorate
  - El Mounira Multiple Sclerosis Unit, Cairo
  - Naser Institute MS Unit, Cairo

IPD SHARING:
Plan to Share IPD: Undecided
It will be only available upon reasonable request from colleagues.